

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Feasibility Study of Ultrasound to Evaluate Muscle-Glycogen Content in Patients with Cancer 2018-1180

| Subtitle: Patient | \$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$\$ |
|---|---|
| Study Chair: Ying Guo | |
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

#### STUDY SUMMARY

The goal of this research study is to learn how well non-invasive MuscleSound<sup>®</sup> technology can be used to learn about levels of glycogen (a type of sugar) in cancer patients during inpatient rehabilitation. The ultrasound information will be processed to represent the energy storage in the muscle. The energy storage in the muscle may help future research to look for dietary plans that can help to increase energy storage, patient exercise tolerance, and functional improvement.

**This is an investigational study.** Future patients may benefit from what is learned. There are no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including potential time commitment or risks. You may not want to participate due to physical activity required.

You can read a full list of potential risks below in the Possible Risks section of this consent.

There is no cost to take part in this study. You may choose not to take part in this study. Your participation in this study can last up to 78 minutes and will be over after you finish Timepoint 3.

#### 1. STUDY DETAILS

# Timepoint 1

If you agree to take part in this study, you will complete questionnaires about your demographic information (such as your sex, age, race), as well as questionnaires about such things as your weight, height, body mass index, medications that you are taking, and your past medical history, diet restrictions, weight loss history in the last 6 months, and the time of your last meal. You will complete a questionnaire about your weight, height, food intake, symptoms, activities and function. These questionnaires (total of 2 pages) should take about 20 minutes to complete.

Your body composition will be recorded by standing on a scale for 1-2 minutes to learn what your body mass index is. This should take about 5 minutes to complete. Using an ultrasound probe and jelly, you will have an ultrasound evaluation of your thigh muscle. Using the image captured, the muscle-glycogen assessment is calculated using an app called MuscleSound<sup>®</sup> technology. MuscleSound<sup>®</sup> will not receive your data or identifiers. The site where the image is taken will be marked, so that 2 more ultrasound images can be taken at the same location during Timepoints 2 and 3. Each ultrasound should take about 3 minutes to complete.

If you are able to complete the ultrasound evaluation, you will immediately move on to Timepoint 2.

# Timepoint 2

You will take part in moderate intensity exercise, which is part of your therapy supervised by your treating therapist, such as cycling or walking for 10 minutes. You will then have an ultrasound evaluation of your thigh muscle again (the same as in Timepoint 1).

If you tolerate this, you will immediately move on to Timepoint 3.

#### Timepoint 3

You will take part in moderate intensity exercise, such as cycling or walking for 10 minutes. You will then have an ultrasound evaluation of your thigh muscle again.

## 2. POSSIBLE RISKS

Mild to moderate **physical activity** may cause sore and/or pulled muscles, heart problems, physical discomfort, and/or accidental injuries such as falling. You may also experience some physical discomfort such as increased heart rate, chest pain, shortness of breath, headache, nausea, and/or fatigue.

The ultrasound probe and jelly may be cold and uncomfortable, but the sensation resolves very quickly afterwards.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen. All study data will be stored in

password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the questionnaires, you are encouraged to contact your doctor or the study chair.

This study may involve unpredictable risks to the participants.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Unless otherwise stated in this consent form, all of the costs linked with this study, which are not covered by other payers (health maintenance organization [HMO], health insurance company, etc.), will be your responsibility.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

## **Additional Information**

- 4. You may ask the study chair (Dr. Ying Guo, at 713-792-6082) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, and you may be asked to sign another informed consent and authorization form stating your continued

willingness to participate in this study.

8. MD Anderson may benefit from your participation and/or what is learned in this study.

#### **Future Research**

Your personal information is being collected as part of this study. This information, or data, may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

Before being shared for future research, every effort will be made to remove your identifying information from any data. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data are used for future research. If this research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data.

# <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

- A. During the course of this study, MD Anderson may be collecting and using your PHI. For legal, ethical, research, and safety-related reasons, the research team may share your PHI with:
  - The Office for Human Research Protections (OHRP)
  - The IRB and officials of MD Anderson
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form
- B. Signing this consent and authorization form is optional but you cannot take part in this study if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible according to state and federal law. However, in some situations, health authorities could be required to reveal the names of participants.

Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.

D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer of MD Anderson at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.

# **CONSENT/AUTHORIZATION**

| I understand the information in this consent form. I have had a characteristic consent form for this study, or have had it read to me. I have had a about it, ask questions, and talk about it with others as needed. I g permission to enroll me on this study. By signing this consent form any of my legal rights. I will be given a signed copy of this consent | chance to think<br>ive the study chair<br>n, I am not giving up |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| LEGALLY AUTHORIZED REPRESENTATIVE (LAR) The following signature line should only be filled out when the part the capacity to legally consent to take part in the study and/or sign or her own behalf. | - |
| SIGNATURE OF LAR | DATE |
| RELATIONSHIP TO PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be performe 2018-1180. | ed under Protocol |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT<br>PRESENTATION (OTHER THAN PHYSICIAN OR STUDY<br>CHAIR) | DATE |
| A witness signature is only required for vulnerable adult participants. If witnessing the assent of a pediatric participant, leave this line blank and sign on the witness to assent page instead. | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his representative, using language that is understandable and appropriate fully informed this participant of the nature of this study and it and risks and that the participant understood this explanation. | riate. I believe that I |
| PERSON OBTAINING CONSENT | DATE |

# I have translated the above informed consent as written (without additions or subtractions) into \_\_\_\_\_\_ and assisted the people \_\_\_\_\_\_ (Name of Language) obtaining and providing consent by translating all questions and responses during the consent process for this participant. NAME OF TRANSLATOR SIGNATURE OF TRANSLATOR DATE □ Please check here if the translator was a member of the research team. (If

checked, a witness, other than the translator, must sign the witness line below.)

SIGNATURE OF WITNESS TO THE VERBAL TRANSLATION (OTHER THAN TRANSLATOR, PARENT/GUARDIAN, OR STUDY CHAIR)

**TRANSLATOR** 

DATE